CLINICAL TRIAL: NCT00165633
Title: A Randomized, Placebo-Controlled, Phase II/III Clinical Study on Inhibitory Effects of E0167 on Recurrence of Hepatocellular Carcinoma
Brief Title: A Phase II/III Clinical Study on Inhibitory Effects of E0167 on Recurrence of Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Customer Information Services Department. CRC and QA, Eisai Company Limited
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E0167-J081-551
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular; Carcinoma; Hepatitis C Virus; Hepatitis B Virus; recurrence; Vitamin K2; E0167
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Hepatitis C; Hepatitis B; Recurrence | interventions — menatetrenone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Menatetrenone
- 2 (Experimental)
  Interventions: Drug: Menatetrenone
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Menatetrenone — 45 mg capsule, orally, three times a day, after meals.
  Other Names: E0167
  Arms: 1
Drug: Menatetrenone — 90 mg capsule, orally, three times a day, after meals.
  Other Names: E0167
  Arms: 2
Drug: Placebo — Placebo capsule, orally, three times a day, after meals.
  Arms: 3

SUMMARY:
The purpose of this study is to determine the superiority of inhibitory effects and safety of Menatetrenone (E0167) on recurrence in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
The study was conducted as a multicenter, randomized, parallel, placebo-controlled, double-blind comparative clinical study. Patients were randomly assigned in a double-blind manner to receive 45 or 90 mg/day of oral vitamin K2 or an identical-appearing placebo. Study drug was administered orally three times daily after meals until recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years or older at the time of obtaining consent.
2. Systemic conditions are 0 to 2 score of Performance Status (according to Eastern Cooperative Oncology Group: ECOG).
3. Diagnosis of hepatocellular carcinoma is based on the following 1) or 2).

   * 1) Patients who are confirmed to have early tumor stain and typical finding(s) of hepatocellular carcinoma with CT or MRI imaging
   * 2) Patients who underwent tumor biopsy and are histopathologically diagnosed as hepatocellular carcinoma
4. Primary onset or recurrence of hepatocellular carcinoma is not more than 1 time.
5. Patients who underwent the following 1) or 2) within 90 days prior to registration to determine therapeutic effect.

   * 1) Patients who underwent local therapy to achieve complete hepatonecrosis and are confirmed to have complete hepatonecrosis with CT imaging or MRI.
   * 2) Patients who underwent surgical treatment(s) and are confirmed not to have residual tumor with CT or MRI imaging.
6. Patients who meet the following items to determine liver function:

   * 1) Albumin is 2.8 g/dL or above
   * 2) Total bilirubin is under 2.0 mg/dL
   * 3) Prothrombin activation is 40% or above
7. Patients who are given full explanation of study participation (including cancer notification) and submit written consent forms with their understanding as well as voluntary will for this study.

Exclusion Criteria:

1. Hepatocellular carcinoma:

   * 1) Patients who have extrahepatic metastasis
   * 2) Patients who have portal invasion
   * 3) Patients who experienced with systemic administration of anti-malignant tumor drugs to treat hepatocellular carcinoma
   * 4) Patients treated with transcatheter arterial chemoembolization (TAE) alone as a non-local therapy for hepatocellular carcinoma
2. Hepatitis:

   -- 1) Patients of (a) or (b) previously treated with interferon preparations (including clinical studies).
   * (a) Patients with chronic hepatitis C virus (HCV) showing HCV-RNA negative
   * (b) Patients with viral hepatitis treated with interferon preparations within the last 2 years (from the same day, 6 months earlier to the day of obtaining consent forms)
   * (c) Patients with encephalopathy in which pharmacotherapy is ineffective
   * (d) Patients with ascites or pleural effusion that cannot be managed with diuretics
3. Systemic conditions:

   * 1) Patients unable to receive oral administration
   * 2) Patients with a history of gastrectomy or extensive resection of digestive tract
   * 3) Patients who are suspected to have biliary occlusion, choleretic disorder, cholecystectomy, or malabsorption of liposoluble agents
   * 4) Patients with complicated serious diseases such as cardiovascular (e.g., myocardial infarction), hematological (e.g., aplastic anemia), and/or renal dysfunctions (e.g., acute and chronic renal failure)
   * 5) Patients with multiple cancers (within a 5-year cancer-free period [from the same day of 5 years earlier to the day of obtaining consent forms])
4. Drug administration:

   * 1) Patients on warfarin potassium therapy
   * 2) Patients with a known history of drug allergy to E0167 or its ingredients
   * 3) Patients who received vitamin K preparations within the recent 6 months (from the same day of 6 month earlier to the day of obtaining consent forms)
5. Other exclusion criteria

   * 1) Women of pregnant, lactating, childbearing potential, or with the intention of becoming pregnant
   * 2) Patients who are presently participating in another clinical study (except for follow-up surveys for study outcomes)
   * 3) Patients who are judged to be ineligible for study entry by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2004-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival period. | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nozomu Koyanagi, Study Director — Eisai Co., Ltd - Development Clinical Research Department. Clinical Research Center
Locations (25):
- Japan (25):
  - Fukuoka, Fukuoka
  - Kurume, Fukuoka
  - Naka, Hiroshima
  - Sapporo, Hokkaido-prefecture
  - Hitachi, Ibaraki
  - Morioka, Iwate
  - Kawasaki, Kanagawa
  - Kanazawa, Kanazawa-prefecture
  - Senndai, Miyagi
  - Niigata, Niigata
  - Ōita, Oita Prefecture
  - Kurashiki, Okayama-ken
  - Okayama, Okayama-ken
  - Moriguchi, Osaka
  - Osaka, Osaka
  - Sayama, Osaka
  - Saga, Saga-ken
  - Shizuoka, Shizuoka
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Wakayama, Wakayama
  - Ube, Yamaguchi